CLINICAL TRIAL: NCT04331886
Title: An Observational Study of Patients With Coronavirus Disease 2019
Acronym: COVID-19
Status: Completed | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-COVID-19
Record Dates: First submitted 2020-03-31; First posted 2020-04-02 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: COVID-19; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study of patients with COVID-19 designed to specifically address important clinical questions that remain incompletely answered for coronavirus disease 2019.

DETAILED DESCRIPTION:
Data from up to 5,000 adult patients in the US will be captured from eligible patients enrolled following admission to the hospital. Participants will have de-identified medical records collected from hospital admission to discharge, including but not limited to critical care monitoring, details on mechanical ventilation, laboratory data, imaging reports, medications, and all procedures. Diagnosis and patient management will follow each hospital's standard of care and no specific treatments, procedures or laboratory tests will be dictated by enrollment in TARGET-COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years) who are or have been hospitalized and diagnosed with Severe Acute Respiratory Syndrome Coronavirus (SARS-CoV-2) infection.
* SARS-CoV-2 confirmed diagnosis (e.g. polymerase chain reaction [PCR] or other clinically utilized test).

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Data for up to 5,000 hospitalized patients with a positive diagnosis of coronavirus disease 2019 (COVID-19) in the United States will be collected in TARGET-COVID-19.
Sampling Method: Non-Probability Sample
Enrollment: 199 (Actual)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-08-20 (Actual); Study Completion 2022-09-26 (Actual)

PRIMARY OUTCOMES:
Natural history of COVID-19: Characteristics of COVID-19 | 12 months
Natural history of COVID-19: Participant demographics | 12 months
Natural history of COVID-19: Treatment use | 12 months
Time point of clinical response | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States